CLINICAL TRIAL: NCT04298190
Title: Dialectical Behavior Therapy vs Enhanced Usual Care for Suicidal and Self-harming Adolescents. Outcomes in Adult Life 10 Years Posttreatment
Brief Title: Dialectical Behavior Therapy vs Enhanced Usual Care for Suicidal and Self-harming Adolescents. 10 Year Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Lars Mehlum, Professor dr med, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ES641048
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Self-Harm, Deliberate; Borderline Personality Disorder
Keywords: self harm; dialectical behaviour therapy; borderline personality disorder; emotional dysregulation
MeSH Terms: conditions — Self-Injurious Behavior; Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialectical Behaviour Therapy (Experimental): Dialectical Behavior Therapy, delivered for 19 weeks, consisted of 1 weekly session of individual therapy (60 minutes), 1 weekly session of multifamily skills training (120 minutes), and family therapy sessions and Telephone coaching with individual therapists outside therapy sessions as needed.
  Interventions: Behavioral: Dialectical Behaviour Therapy for Adolescents (DBT-A)
- Enhanced Usual Care (Active Comparator): Enhanced usual care was 19 weeks of standard care (enhanced for the purpose of the study by requiring that EUC therapists agree to provide on average no less than 1 weekly treatment session per patient throughout the trial) delivered by therapists (4 psychiatrists, 16 clinical psychologists, 6 clinical social workers, 2 clinical pedagogues, 1 specialist nurse, and 1 psychology graduate student) not trained in or practicing DBT.
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: Dialectical Behaviour Therapy for Adolescents (DBT-A) — 16 weeks of Dialectical behavior therapy with one weekly session of individual therapy, one weekly session of multifamily skills training group, telephone coaching and ancillary family therapy and/or pharmacological treatment as needed.
  The treatment has been developed by Marsha Linehan (Linehan, 1993a; 1993b)and adapted for adolescents by Alec Miller (Miller, Rathus & Linehan, 2007). Individual DBT therapists have been trained by drs Alec L Miller and Sarah K Reynolds and have a minimum of one year clinical practise as DBT therapists. The therapists are organised in two consultation teams supervised on a bimonthly basis throughout the entire study by drs Miller and Reynolds respectively.
  Arms: Dialectical Behaviour Therapy
Behavioral: Enhanced usual care — 16 weeks of outpatient treatment in child and adolescent psychiatric clinics in Oslo, on average one weekly session of individual therapy and ancillary supportive family and/or pharmacological treatment as needed.
  Arms: Enhanced Usual Care

SUMMARY:
The purpose of the study is to evaluate the long-term efficacy of dialectical behavior therapy (DBT) in treatment of adolescents with deliberate self harm compared to enhanced usual care (EUC). This study follows-up 77 patients in the ages of 12-18 yrs who have been included in an RCT of DBT-A vs EUC. The main inclusion criterion for this study was repetitive self-harm behaviour. The patients were randomly allocated to receive 16 weeks of outpatient DBT or EUC in child and adolescent psychiatric clinics in Oslo. Participants have been assessed so far on six different time-points: baseline (before starting treatment), 9 weeks, 15 weeks, 19 weeks, 71 weeks and 3 years after start of the treatment. In the current project patients will be assessed a 7th time 10 years after treatment completion.

It is hypothesized that compared with participants who had received EUC in the original trial during their adolescence participants who had received DBT-A will:

A) report a significantly lower frequency of episodes of self-harm, both last year and over the extended 10-year follow-up interval.

B) be significantly less impaired with respect to social, family and occupational functioning and report a higher quality of life.

C) have retained significantly fewer diagnostic criteria of BPD and have less severe borderline features according to dimensional measures and have significantly fewer signs of emotion dysregulation.

DETAILED DESCRIPTION:
Suicide attempts and non-suicidal self-harm, highly prevalent in adolescents, are behaviours strongly associated with severe emotion dysregulation, mental health problems and increased suicide risk. The original study, on which the present study is building, used a randomized controlled design, with a stratified block randomization procedure, and blinded pre-treatment, post-treatment and follow-up evaluations comparing 19weeks of DBT-A with EUC of equal length.

Of special interest to this follow-up study is to gain more knowledge on their capacity to regulate emotions, since failures in emotion regulation is an underlying mechanism of repetitive self-harm behaviours and several other difficulties, and since a main aim of DBT-A is to enhance adolescents capacity to use healthy emotion regulation strategies. The study is designed to carefully include user and family perspectives on the definition of specific outcomes and how to measure them, we will collect detailed data on important outcomes employing a combination of quantitative and qualitative methods, innovative approaches such as ecological momentary assessment and register data. Adding new data to the existing rich data will give us a basis to study the dynamic interplay between symptoms, emotions, and functional and dysfunctional behaviours and make new discoveries of mechanisms of therapeutic change, knowledge to further increase treatment response rates and individualize treatments and to inform further development of this treatment and its implementation in Norway and other countries.

The proposed study will investigate:

1. the 10-year post-randomization treatment outcomes of DBT-A compared with EUC with respect to: a) frequency of subsequent episodes of self-harm, b) severity of suicidal ideation, c) level of depressive symptoms and d) frequency of subsequent emergency room visits, hospitalizations and use of additional treatments due to risk of self-harm behaviour.
2. the 10-year post-randomization clinical course and stability of a diagnosis of BPD, its diagnostic criteria and borderline symptoms.
3. participants' adult mental health, social, family and occupational functioning and quality of life.
4. participants' adult strategies for and capacity to cope with stressful life-events and situations in their daily lives and effectively regulate emotions.
5. the association between participants' adult life use of skills and functional coping strategies and self-harm behaviour and other problem behaviours, and whether any substitution from onedysfunctional coping behaviour to another has occurred.
6. participants' evaluation of what components of the treatment was most helpful and led to the strongest and most persistent change in important functions and aspects of life.
7. the economic cost of treatments consumed and functional impairment and occupational disability over the 10-year post-randomization period and the long-term cost-effectiveness of DBT-A.

ELIGIBILITY:
The inclusion criteria for the initial study were:

1. History of repeated self-harm (last episode within last 4 months) and
2. Age between 12 and 18 years and
3. Satisfied at least 2 criteria of DSM-IV Borderline Personality Disorder (BPD) (as measured by the SCIDII) (in addition to the self-destructive criterion) - alternatively at least 1 criterion of DSM-IV BPD plus at least 2 threshold level criteria and
4. Written informed consent from patient and parent(s) to participate in the study and
5. Patient fluently Norwegian speaking

Exclusion Criteria:

1. Psychotic disorders or
2. Anorexia nervosa or
3. Severe substance dependence disorders or
4. Mental retardation (IQ less than 70) or
5. Asperger syndrome/autism -

Ages: 22 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Frequency of subsequent episodes of self-harm | 10 years
  Measured by the Linehan Parasuicide Count (LPC)

SECONDARY OUTCOMES:
Severity of suicidal ideation | 10 years
  Measured by the Suicidal Ideation Questionnaire Jr (SIQ-Jr). Scale range: min= 0, max = 90. High values represent a worse outcome.
Self-reported evel of depressive symptoms | 10 years
  Measured by the Moods and feelings questionnaire (MFQ). Scale range: min = 0, max = 26. High levels represent a worse outcome
Researcher rated level of depressive symptoms | 10 years
  Measured by the Montgomery Asberg Depression Rating Scale (MADRS). Scale range: min=0, max=60. High levels represent a worse outcome
Frequency of subsequent emergency room visits, hospitalizations and use of additional treatments due to risk of self-harm behaviour | 10 years
  Measured through and interview specifically developed for the purpose and through linkage with the Norwegian Patient Register

CONTACTS AND LOCATIONS:
Overall Officials: Lars Mehlum, MD PhD, Principal Investigator — University of Oslo
Locations (1):
- National Centre for Suicide Research and Prevention Unit/University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linehan, M.M. (1993a). Cognitive-behavioral treatment of borderline personality disorder. New York: Guilford Press
- [Background] Linehan, M.M. (1993b). Skills training manual for treating borderline personality disorder. New York: Guilford Press
- [Background] Miller, A.L., Rathus J.H., Linehan, M.M. (2007). Dialectical behavioral therapy with suicidal adolescents. New York: Guilford Press
- [Derived] Mehlum L, Dibaj IS, Haga E, Helle SE, Morken KTE, Klungsoyr O, Tormoen AJ. Adult life outcomes for adolescents 12.4 years after dialectical behavior therapy - a randomized clinical trial. Eur Child Adolesc Psychiatry. 2026 Jan 16. doi: 10.1007/s00787-025-02856-w. Online ahead of print. PMID 41543545
- See also: Information about the research project in Norwegian — http://www.med.uio.no/klinmed/forskning/sentre/nssf/forskning/nssf-prosjekter/dbt-langtidseffekt/